CLINICAL TRIAL: NCT02759627
Title: Does Isolated Robotic-Assisted Gait Training Improve Functional Status, Daily Living And Quality Of Life In Stroke Patients?: A Single-Blinded Randomized Controlled Study
Brief Title: Does Isolated Robotic-Assisted Gait Training Improve Functional Status, Daily Living And Quality Of Life In Stroke?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, RUSTEM MUSTAFAOGLU, MSc, PT, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-22
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Cerebrovascular Stroke; Cerebrovascular Accident; Cerebral Stroke
Keywords: Rehabilitation; Gait; Ambulation; Exercise Therapy; Physical Exertion; Motor Skills
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional Training (No Intervention): Conventional physical therapy consisted of neurophysiological concepts such as Bobath and Brunnstrom.Training sessions focused on static and dynamic postural tasks, improving lower and upper extremity range of motion, strengthening and overground walking. During walking training, emphasis was on distance walked than on gait quality. Symmetrical weight distribution was encouraged through verbal and tactile cues and was made more difficult by the addition of arm activities or actions requiring trunk rotation. In an effort to improve rhythmic weight-shifting ability, subjects practiced shifting their weight in forward and backward directions and side to side while performing reaching tasks. A session lasted 45 minutes, for 5 days per week for 6 weeks.
- Robotic-Assisted Gait Training (Experimental): Lokomat (Hocoma) was used in Robotic-Assisted Gait Training group with 20 % body weight reduced. The participants walked on device at 1.8 km/h (0.5 m/sec) velocity. For each participant body weight portion was ensured by a security belt while walking. Each session took 45 minutes including setup, commands and rest time. Verbal instructions were used for encouragement but no manual assistance was given to improve gait. Robotic-Assisted Gait Training sessions lasted 45-minute sessions, 2 days a week during 6 weeks.
  Interventions: Other: Robotic-Assisted Gait Training
- Combined Training (No Intervention): Combined Training consisted of inpatient participants who were treated with 45 minute-conventional training, 5 days a week during 6 weeks. Additionally this group had 45 minute-Robotic-Assisted Gait Training, 2 days a week during 6 weeks.

INTERVENTIONS:
Other: Robotic-Assisted Gait Training — There were three intervention arms in this study,
  1. Robotic-Assisted Gait Training,
  2. Conventional Training,
  3. Combined Training.
  Arms: Robotic-Assisted Gait Training

SUMMARY:
Stroke is one of the major cause of morbidity and mortality and the leading cause of disability in adults all around the world. Stroke survivors can suffer several neurological impairments and deficits which have an important impact on patient's quality of life and which increase the costs for health and social services. After stroke, impairments in ADLs and functional status, deterioration in health related quality of life can be seen.

Although most of the stroke survivors experience some level of neurological recovery, nearly 50%-60% of stroke patients still experience some degree of motor impairment, and approximately 50% are at least partly dependent in activities-of-daily-living (ADL). Gait recovery, performing activities of daily living and regaining independence in ADLs are the main focus of stroke rehabilitation programs.

Robotic technologies are becoming more promising techniques for the locomotor training in stroke patients. Achieving a functional walking level is one of the target of robotic gait training and it has been shown that Robotic-Assisted Gait Training (RAGT) improves walking function in stroke patients. Having a functional gait level may help the stroke patients to regain independence in ADLs and improve quality of life.

The purpose of the present study was to investigate the effects of RAGT on functional status, ADLs and health related quality of life.

DETAILED DESCRIPTION:
Design:

Our study design was a randomized single-blind controlled study of 6 weeks including inpatient ambulatory subacute and chronic stroke patients. Sample size was calculated by Raosoft, Inc. Clinically meaningful difference was considered 20% for all outcome measures. The original sample size was estimated 45 patients to detect a statistically significant difference between groups. Considering the drop-out, fifty-one patient were included. The patients were randomly assigned to one of three training group by a researcher (ARO) using the function of Microsoft Office Excel software.

In this randomized-controlled study, eighty patients were assessed in terms of eligibility criteria, and 51 patients were included in the study. The patients were evaluated by two physiatrists in Istanbul Physical Medicine and Rehabilitation Education and Research Hospital and referred to the Physiotherapy and Rehabilitation Unit of the same hospital. Enrollment period was between November 2014 and December 2015.

Blinding:

During the consent process, participants were advised that they would be randomized to one of three intervention groups. To minimize exposure between groups, the Robot-Assisted Gait Training and Conventional Training programs were administered in different sections of the rehabilitation center. The 2 trial physiotherapists could blinded to intervention group. All treatment schedules were planned by another researcher. All outcome assessments were conducted by a blinded assessor located offsite. Trial staff instructed participants to avoid mentioning anything about their intervention to the assessor. Patients were asked not to shear any information about treatment between each other.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of a stroke (at least 3 months),
* ambulatory with or without the use of an assistive device or ankle-foot orthosis,
* 3 or higher grades in Functional Ambulation Category,
* able to walk 10 meters with or without supervision,
* able to follow verbal instructions,
* physician approval to enter an exercise program.

Exclusion criteria:

* previous stroke history,
* any other neurologic disorders, complications from other health conditions (cardiovascular or musculoskeletal conditions),
* contracture or muscle tonus ≥ 3 according to Modified Ashworth Scale, preventing range of motion in lower extremity,
* severe osteoporosis,
* cognitive deficit preventing them from following instructions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The Barthel Index (BI) | 6 weeks
  The BI was used to determine the level of independence in functional activities and included ten items. The score ranges from 0-100, and a higher BI score indicates better functioning. Minimal clinically important difference for BI is 18.5 points.
The Stroke Specific Quality of Life Scale (SSQOL). | 6 weeks
  The Stroke Specific Quality of Life scale (SS-QOL) was used to address the ICF participation component.The score for the questionnaire is between 26 (lowest social participation) and 130 (highest social participation).
The 6-Minute Walk Test (6MWT) | 6 weeks
  Walking function was assessed by distance walked in 6 minutes (6MWT).Usual ambulatory devices, lower-extremity orthotics, and stand-by assistance were permitted. Therapists closely guarded participants during gait testing, but did not provide physical assistance. For the 6-minute walk test, participants walked through continuous hallways with minimal foot traffic. End of the test walked distance recorded by meter.
The Stair Climbing ascend and descend tests (SCas and SCde) | 6 weeks
  Participants climbed up and down 10 steps (measuring 18 cm in height), with or without the use of the rails and/or assistive devices. Subjects were asked to climb the stairs without skipping any steps, preferably using one foot for each step and descend without stopping. The time taken to climb up and down the 10 steps was recorded as a second.

SECONDARY OUTCOMES:
The Fugl-Meyer Assessment (FMA) | 6 weeks
  Lower limb impairment and balance were measured by Fugl-Meyer Lower Extremity Assessment (FMA-LE).FMA-LE consists of 17 items, with a maximum possible score of 34 points. Each item was answered using a 3-point ordinal scale (0 = cannot perform, 1 = can partially perform, 2 = can fully perform).
The Comfortable 10-m Walk Test (CWT) | 6 weeks
  CWT was used to determine the speed of comfortable walking. The test was applied in a 14 meter-corridor. The patients were wanted to walk comfort and allowed to use walking aid. At 2nd meter the stopwatch was started and stopped when the patient reached the 12th meter. After three trials the average of the three trials was recorded as a second.
Rate of Perceived Exertion (RPE) | 6 weeks
  Rate of Perceived Exertion was assessed at the end of 6 MWT and the patients were asked to identify their level of exertion between 6-20.All measurements of were performed before the intervention (baseline) and after the intervention (post treatment).
The Fast 10-m Walk Test (FWT) | 6 weeks
  FWT was used to determine the speed of fast walking. The test was applied in a 14 meter-corridor. The patients were wanted to walk fast and allowed to use walking aid. At 2nd meter the stopwatch was started and stopped when the patient reached the 12th meter. After three trials the average of the three trials was recorded as a second.

CONTACTS AND LOCATIONS:
Overall Officials: IPEK YELDAN, Assoc.prof, Study Director — Istanbul University, Faculty of Health Sciences, Division of Physiotherapy and Rehabilitation Istanbul, Turkey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belda-Lois JM, Mena-del Horno S, Bermejo-Bosch I, Moreno JC, Pons JL, Farina D, Iosa M, Molinari M, Tamburella F, Ramos A, Caria A, Solis-Escalante T, Brunner C, Rea M. Rehabilitation of gait after stroke: a review towards a top-down approach. J Neuroeng Rehabil. 2011 Dec 13;8:66. doi: 10.1186/1743-0003-8-66. PMID 22165907
- [Background] Dombovy ML, Basford JR, Whisnant JP, Bergstralh EJ. Disability and use of rehabilitation services following stroke in Rochester, Minnesota, 1975-1979. Stroke. 1987 Sep-Oct;18(5):830-6. doi: 10.1161/01.str.18.5.830. PMID 3629639
- [Background] Schaechter JD. Motor rehabilitation and brain plasticity after hemiparetic stroke. Prog Neurobiol. 2004 May;73(1):61-72. doi: 10.1016/j.pneurobio.2004.04.001. PMID 15193779
- [Background] Mao YR, Lo WL, Lin Q, Li L, Xiao X, Raghavan P, Huang DF. The Effect of Body Weight Support Treadmill Training on Gait Recovery, Proximal Lower Limb Motor Pattern, and Balance in Patients with Subacute Stroke. Biomed Res Int. 2015;2015:175719. doi: 10.1155/2015/175719. Epub 2015 Nov 16. PMID 26649295
- [Background] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Green J, Forster A, Young J. A test-retest reliability study of the Barthel Index, the Rivermead Mobility Index, the Nottingham Extended Activities of Daily Living Scale and the Frenchay Activities Index in stroke patients. Disabil Rehabil. 2001 Oct 15;23(15):670-6. doi: 10.1080/09638280110045382. PMID 11720117
- [Background] Silva SM, Correa FI, Faria CD, Correa JC. Comparison of quality-of-life instruments for assessing the participation after stroke based on the International Classification of Functioning, Disability and Health (ICF). Braz J Phys Ther. 2013 Sep-Oct;17(5):470-8. doi: 10.1590/S1413-35552012005000118. Epub 2013 Oct 21. English, Portuguese. PMID 24173349
- [Background] Silva SM, Correa FI, Faria CD, Correa JC. Psychometric properties of the stroke specific quality of life scale for the assessment of participation in stroke survivors using the rasch model: a preliminary study. J Phys Ther Sci. 2015 Feb;27(2):389-92. doi: 10.1589/jpts.27.389. Epub 2015 Feb 17. PMID 25729175
- [Background] Lennon S, Baxter D, Ashburn A. Physiotherapy based on the Bobath concept in stroke rehabilitation: a survey within the UK. Disabil Rehabil. 2001 Apr 15;23(6):254-62. doi: 10.1080/096382801750110892. PMID 11336098
- [Background] Visintin M, Barbeau H. The effects of body weight support on the locomotor pattern of spastic paretic patients. Can J Neurol Sci. 1989 Aug;16(3):315-25. doi: 10.1017/s0317167100029152. PMID 2766124
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Hsieh YW, Wang CH, Wu SC, Chen PC, Sheu CF, Hsieh CL. Establishing the minimal clinically important difference of the Barthel Index in stroke patients. Neurorehabil Neural Repair. 2007 May-Jun;21(3):233-8. doi: 10.1177/1545968306294729. Epub 2007 Mar 9. PMID 17351082
- [Derived] Mustafaoglu R, Demir R, Demirci AC, Yigit Z. Effects of core stabilization exercises on pulmonary function, respiratory muscle strength, and functional capacity in adolescents with substance use disorder: Randomized controlled trial. Pediatr Pulmonol. 2019 Jul;54(7):1002-1011. doi: 10.1002/ppul.24330. Epub 2019 Apr 26. PMID 31026384